CLINICAL TRIAL: NCT06481137
Title: InvesTigAtion of the reVersIbility of caRdiac Conduction disturbancEs Following Percutaneous Aortic ValvE Implantation in Patients With Severe aoRtic StEnosis: The TAVI-REVERSE Study
Brief Title: Reversibility of Cardiac Conduction Disturbances Following TAVI
Acronym: TAVI-REVERSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Hospital Universitario La Paz (Other); Hospital Vall d'Hebron (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario A Coruna Spain (Unknown); Hospital Clinico Universitario de Santiago (Other); Hospital Universitario Central de Asturias (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Guillem Muntané Carol, Principal Investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ICPS025/24; PI23/00310 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2024-06-19; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Aortic Stenosis; Transcatheter Aortic Valve Implantation; Conduction Disturbances
Keywords: Aortic stenosis; Transcatheter Aortic Valve Implantation; Conduction Disturbances
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive initial (3-7 days following TAVI) electrophysiological study (EP+) (Experimental): Permanent pacemaker implantation. Continuous ECG monitoring during 4 weeks. Second EP study 30-45 days after TAVI.
  Interventions: Diagnostic Test: Electrophysiological study (EP study); Diagnostic Test: ePatch (extended Holter Monitoring)
- Negative initial (3-7 days following TAVI) electrophysiological study (EP-) (Other): Continuous ECG monitoring during 4 weeks.
  Interventions: Diagnostic Test: ePatch (extended Holter Monitoring)

INTERVENTIONS:
Diagnostic Test: Electrophysiological study (EP study) — Electrophysiological study: A second EP study 30-45 days after TAVI will be performed in the group of patients with positive EP study 3-7 days after TAVI.
  Arms: Positive initial (3-7 days following TAVI) electrophysiological study (EP+)
Diagnostic Test: ePatch (extended Holter Monitoring) — Continuous cardiac rhythm monitoring using the ePatch (Philips) will be performed during 4 weeks after TAVI

SUMMARY:
The management of patients with conduction disturbances (CDs) after transcatheter aortic valve implantation (TAVI) is unclear, especially in those with de novo electrocardiographic CDs (ECG-CDs) such as left bundle branch block.

In this study, the investigators will evaluate the incidence of retrogradation of infra-Hisian CDs in patients with de novo ECG-CDs and positive electrophysiological study (EPS) 3-7 days following TAVI. In addition, the investigators will evaluate the need for cardiac pacing and the incidence of clinical events in patients with negative EPS performed 3-7 days following TAVI.

In this multicenter, longitudinal, prospective study, patients with clinical indication of EP study due to new-onset ECG-CDs after TAVI will be included. A permanent pacemaker will be implanted in patients with positive EPS and a second EPS will be performed in 30-45 days. Additionally, these patients will undergo 4-week continuous monitoring using the ePatch (Philips) long-term Holter recorder, to identify episodes of paroxysmal complete atrioventricular block. Patients with negative EP study will undergo clinical follow-up and continuous monitoring for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for electrophysiological (EP) study after TAVI implantation according to European Guidelines. Patients must have persistent electrocardiographic conduction disturbances (ECG-CDs) that are present from day 2 after TAVI implantation (≥ 48h post-procedure):
* De novo LBBB with QRS complex >150ms and/or PR interval ≥240ms.
* QRS widening or post-procedural PR lengthening > 20ms in patients with baseline ECG-CDs.

Exclusion Criteria:

* Patients with previous pacemaker or implantable defibrillator.
* Patients with baseline complete right bundle branch block.
* Patients in need of cardiac resynchronization or physiological stimulation following TAVI.
* Valve-in-valve procedures.
* TAVI procedures in patients with severe aortic insufficiency.
* Inability to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of retrogradation | 30 days
  1. Patients with positive EP: Evaluate the incidence of retrogradation of infra-Hisian conduction disturbance at 30-45 days following TAVI.
Need for cardiac pacing (incidence of advanced atrioventricular block) | 30 days
  2. Patients with negative EP: Evaluate the rate of patients in need for cardiac pacing (incidence of clinical events related to advanced atrioventricular block).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study procotol and ICF will be shared trough PI request during the duration of the study
Supporting Information: Study Protocol, ICF
Time Frame: During the duration of the study
Access Criteria: Request to the PI